CLINICAL TRIAL: NCT05014412
Title: A PHASE 1/2, OPEN-LABEL, MULTICENTER STUDY TO EVALUATE A DOSING REGIMEN WITH TWO STEP-UP PRIMING DOSES AND LONGER DOSING INTERVALS OF ELRANATAMAB (PF-06863135) MONOTHERAPY IN PARTICIPANTS WITH RELAPSED/REFRACTORY MULTIPLE MYELOMA
Brief Title: A Study to Learn About the Study Medicine (Elranatamab) in Participants With Multiple Myeloma That Has Come Back After Responding to Treatment or Has Not Responded to Treatment
Acronym: MagnetisMM-9
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C1071009; MagnetisMM-9 (Other: Alias Study Number)
Record Dates: First submitted 2021-08-03; First posted 2021-08-20 (Actual); Results first posted 2024-07-30 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
Keywords: BCMA; Multiple Myeloma; Relapse/Refractory; RRMM; Elranatamab; Targeted T-cell; MagnetisMM; MM9; Phase 2; B-Cell Maturation Antigen; monoclonal antibody
MeSH Terms: conditions — Multiple Myeloma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1 (Experimental): Evaluation of step-up priming dosing
  Interventions: Drug: Elranatamab
- Part 2A (Experimental): Dose determination
  Interventions: Drug: Elranatamab
- Part 2B (Experimental): Dose expansion
  Interventions: Drug: Elranatamab
- Part 2C (Experimental): To explore higher dose intensity
  Interventions: Drug: Elranatamab

INTERVENTIONS:
Drug: Elranatamab — BCMA-CD3 bispecific antibody

SUMMARY:
The purpose of the study (Part 1 and Part 2) is to evaluate the safety of a step-up dosing approach (starting with low doses followed by higher doses) of the study medicine (elranatamab) in participants with multiple myeloma that has come back after responding to treatment or has not responded to treatment (relapsed/refractory multiple myeloma). This study will also look at the safety and efficacy of different doses of elranatamab, as well as different intervals between doses.

Participants in the study will receive elranatamab as an injection under the skin at the study clinic. After the initial step-up doses, participants will start receiving one dose every week. The frequency of clinic visits for injections may then decrease over time. Participation will be at least two years.

DETAILED DESCRIPTION:
The purpose of the study (Part 1 and Part 2) of the study is to evaluate the safety (in particular the rate of Grade ≥ 2 CRS) of a step-up priming dose regimen of elranatamab in participants with relapsed/refractory multiple myeloma. In addition, this study will assess the safety of different dosing regimens of elranatamab and if it can provide a clinical benefit in those participants. Elranatamab is a bispecific antibody: binding of elranatamab to CD3-expressing T-cells and BCMA-expressing multiple myeloma cells causes targeted T-cell-mediated cytotoxicity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma (IMWG criteria, Rajkumar et al, 2014)
* Measurable disease, as defined by at least 1 of the following:

  1. Serum M-protein >0.5 g/dL by SPEP
  2. Urinary M-protein excretion >200 mg/24 hours by UPEP
  3. Serum immunoglobulin FLC≥10 mg/dL (≥100 mg/L) AND abnormal serum immunoglobulin kappa to lambda FLC ratio
* Refractory to at least one IMiD
* Refractory to at least one PI
* Refractory to at least one anti-CD38 antibody
* Relapsed/refractory to last anti-myeloma regimen
* ECOG performance status ≤1
* Resolved acute effects of any prior therapy to baseline severity or CTCAE Grade ≤1
* Not pregnant and willing to use contraception

Exclusion Criteria:

* Smoldering multiple myeloma
* Active Plasma cell leukemia
* POEMS syndrome
* Amyloidosis
* Waldenström's macroglobulinemia
* Known active CNS involvement or clinical signs of myelomatous meningeal involvement
* Stem cell transplant within 12 weeks prior to enrollment or active GVHD
* Active HBV, HCV, SARS-CoV2, HIV, or any active, uncontrolled bacterial, fungal, or viral infection
* Any other active malignancy within 3 years prior to enrollment, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ or Stage 0/1 malignancy with minimal risk of recurrence per investigator.
* Previous treatment with an anti-BCMA bispecific antibody or CAR-T cell therapy.
* Live attenuated vaccine within 4 weeks of the first dose
* Previous administration with an investigational drug within 30 days or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer)
* Known or suspected hypersensitivity to the study intervention, or any of its excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2025-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (50):
- United States (35):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care & Hematology - Fort Collins, Fort Collins, Colorado
  - Poudre Valley Health System (PVHS), Fort Collins, Colorado
  - UCHealth Cancer Care & Hematology - Greeley, Greeley, Colorado
  - UCHealth Cancer Care & Hematology - Loveland, Loveland, Colorado
  - UF Health Shands Cancer Hospital, Gainesville, Florida
  - UF Health Shands Hospital Pharmacy Investigational Drug Service - Main, Gainesville, Florida
  - UF Health Shands Hospital, Gainesville, Florida
  - East Jefferson General Hospital Bone Marrow Transplant Clinic, Metairie, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - Tulane University, New Orleans, Louisiana
  - The Regents of the University of Michigan, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - MSK Basking Ridge, Basking Ridge, New Jersey
  - MSK Monmouth, Middletown, New Jersey
  - MSK Bergen, Montvale, New Jersey
  - MSK Commack, Commack, New York
  - MSK Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center - Investigational Drug Service Pharmacy, Long Island City, New York
  - Memorial Sloan Kettering Cancer Center - David H. Koch Center for Cancer Care (74th Street)., New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MSK Nassau, Uniondale, New York
  - Cleveland Clinic Taussig Cancer Institute, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - St. David's South Austin Medical Center, Austin, Texas
  - Texas Oncology-South Austin, Austin, Texas
  - Blood Cancer and Stem Cell Transplant Clinic, San Antonio, Texas
  - Methodist Healthcare System of San Antonio dba Methodist Hospital, San Antonio, Texas
  - Methodist Hospital Investigational Pharmacy, San Antonio, Texas
  - Methodist Plaza Clinical Trials Office, San Antonio, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
  - University of Utah, Salt Lake City, Utah
- Japan (5):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Japanese Red Cross Medical Center, Shibuya-ku, Tokyo
  - University Hospital,Kyoto Prefectural University of Medicine, Kyoto
- Taiwan (3):
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (7):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - University College London Hospitals NHS Foundation Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - King's College Hospital NHS Foundation Trust, London
  - The Royal Marsden NHS Foundation Trust, London
  - University College London Hospitals NHS Foundation Trust NIHR, London
  - The Royal Marsden NHS Foundation Trust, Surrey

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Lon HK, Hibma J, Jiang S, Sullivan S, Vandendries E, Skoura A, Wang D, Elmeliegy M. Population Exposure-Response Efficacy Analysis of Elranatamab (PF-06863135) in Patients with Multiple Myeloma. Target Oncol. 2025 Sep;20(5):803-819. doi: 10.1007/s11523-025-01168-y. Epub 2025 Aug 18. PMID 40826257
- [Derived] Elmeliegy M, Viqueira A, Vandendries E, Hickman A, Conte U, Irby D, Hibma J, Lon HK, Piscitelli J, Soltantabar P, Skoura A, Jiang S, Wang D. Dose Optimization of Elranatamab to Mitigate the Risk of Cytokine Release Syndrome in Patients with Multiple Myeloma. Target Oncol. 2025 Mar;20(2):349-359. doi: 10.1007/s11523-025-01134-8. Epub 2025 Feb 25. PMID 40000533
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1071009

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this study Part 2C was exploratory and there was no participant enrolled in Part 2C as it was not conducted. A total of 86 participants with relapsed/ refractory multiple myeloma were enrolled in this study and 85 participants were treated.
Pre-assignment Details: Results are reported only for primary outcome measure and those secondary outcome measures whose analysis was final at primary completion date (15-June-2023). Remaining secondary outcome measures results would be reported once analysis is final.
Groups:
- Part 1: Participants received elranatamab 4 milligram (mg) on Cycle (C) 1 Day 1 (D) [C1D1] and 20 mg on C1D4 and then 76 mg every week (QW) for 6 cycles. Thereafter, participants with partial response (PR) or better response persisting for greater than equal to (>=) 2 months on QW received 76 mg every 2 weeks (Q2W) and/or 116 mg or 152 mg every 4 weeks (Q4W) from C7 and onwards. One cycle =28 days. Treatment continued until confirmed disease progression, unacceptable toxicity, withdrawal of consent, or study termination.
- Part 2A: Dose Level 1: Participants received elranatamab 4 mg on C1D1 and 20 mg on C1D4 and then 76 mg QW for 1 cycle. Thereafter, in dose level 1 received 116 mg Q2W for C2 to C6 and 116 mg Q4W from C7 and onwards (participants with PR or better response persisting for >= 2 months on Q2W). One cycle =28 days. Treatment continued until confirmed disease progression, unacceptable toxicity, withdrawal of consent, or study termination.
- Part 2A: Dose Level 2: Participants received elranatamab 4 mg on C1D1 and 20 mg on C1D4 and then 76 mg QW for 1 cycle. Thereafter, in dose level 2 participants received 152 mg Q2W for C2 to C6 and 152 mg Q4W from C7 and onwards (participants with PR or better response persisting for >= 2 months on Q2W). One cycle =28 days. Treatment continued until confirmed disease progression, unacceptable toxicity, withdrawal of consent, or study termination.
- Part 2B: Participants received elranatamab 4 mg on C1D1 and 20 mg on C1D4 and then 76 mg QW for 1 cycle. Thereafter, participants were received 116 or 152 mg Q2W for C2 to 6 and 116 mg or 152 mg Q4W from C7 and onwards (participants with PR or better response persisting for >=2 months on Q2W). One cycle =28 days. Treatment continued until confirmed disease progression, unacceptable toxicity, withdrawal of consent, or study termination.
Period: Overall Study
Arm/Group | Part 1 | Part 2A: Dose Level 1 | Part 2A: Dose Level 2 | Part 2B
Started | 33 | 12 | 11 | 29
Completed | 0 | 0 | 0 | 0
Not Completed | 33 | 12 | 11 | 29
Not completed — Death | 11 | 7 | 4 | 7
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 2
Not completed — Ongoing | 21 | 4 | 6 | 20

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 dose of study intervention.
Groups:
- Part 1: Participants received elranatamab 4 mg on C1D1 and 20 mg on C1D4 and then 76 mg QW for 6 cycles. Thereafter, participants with PR or better response persisting for >= 2 months on QW received 76 mg every Q2W and/or 116 mg or 152 mg Q4W from C7 and onwards. One cycle =28 days. Treatment continued until confirmed disease progression, unacceptable toxicity, withdrawal of consent, or study termination.
- Total: Total of all reporting groups
Arm/Group | Part 1 | Part 2A: Dose Level 1 | Part 2A: Dose Level 2 | Part 2B | Total
Number analyzed (Participants) | 33 | 12 | 11 | 29 | 85
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.4 (10.14) | 64.0 (8.75) | 66.8 (11.12) | 64.1 (8.08) | 63.0 (9.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 4 | 5 | 15 | 43
  Male | 14 | 8 | 6 | 14 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 2 | 5
  Not Hispanic or Latino | 30 | 12 | 9 | 22 | 73
  Unknown or Not Reported | 1 | 0 | 1 | 5 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 19 | 5 | 3 | 8 | 35
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 1 | 4
  White | 11 | 6 | 7 | 17 | 41
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 2 or Higher Cytokine Release Syndrome (CRS) During Cycle 1: Parts 1 and 2
Description: CRS: supraphysiologic response following any immune therapy that results in the activation or engagement of endogenous or infused T-cells and/or other immune effector cells. Symptoms must include fever at the onset, and may include hypotension, hypoxia and end organ dysfunction. As per ASTCT criteria, Grade (G) 1: fever (temperature >=38 degree Celsius), hypotension and/or hypoxia none; G 2: fever, hypotension not requiring vasopressors, hypoxia requiring low-flow nasal cannula/ facemask or blow-by; G 3: fever, hypotension requiring a vasopressor with or without vasopressin, hypoxia requiring high-flow nasal cannula/ facemask, nonrebreather mask, or Venturi mask; G 4: fever, hypotension requiring multiple vasopressors (excluding vasopressin), hypoxia requiring positive pressure. Organ toxicities associated with CRS graded according to CTCAE v5.0. G 1: Mild, G 2: Moderate, G 3: severe, and G 4: life-threatening consequences; urgent intervention indicated. G 5: death related to AE.
Time Frame: Parts 1 and 2: Cycle 1 (28 days)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study intervention. Data for this outcome is presented for all participants in Part 1 and 2 of the study (combined) per study design, as all treatment groups utilized the same elranatamab priming regimen (4 mg on Day 1/20 mg on Day 4, followed by 76mg QW) during Cycle 1.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: All participants who were enrolled and treated in Part 1 and 2 of the study and evaluated for CRS.
Arm/Group | All Participants
Number analyzed (Participants) | 85
Participants | 12

2. Secondary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs): Part 2A
Description: Hematological: grade 4 neutropenia lasting >5 days; febrile neutropenia; grade >=3 neutropenia with infection; grade 4 thrombocytopenia; grade 3 thrombocytopenia with grade >=2 bleeding. Non-hematological: grade >=4 adverse events (AEs); grade 3 CRS (except CRS events: not been maximally treated or improved to grade <=1 within 48 hours); grade 3 AEs (except: AEs attributed to a CRS event; grade 3 nausea, vomiting and diarrhea that improve to grade <= 2 within 72 hours after maximal medical management has been initiated, grade 3 fatigue lasting <1 week; grade 3 AEs that recover to baseline or grade 1 within 5 days); confirmed drug-induced liver injury meeting Hy's law criteria; grade 3-4 laboratory abnormalities; other clinically important or persistent AEs; Grade 3 injection site reaction. CTCAE version 5.0: Grade 1: Mild AE, Grade 2: Moderate, Grade 3: severe, and grade 4: life-threatening consequences; urgent intervention indicated. Grade 5: death related to AE.
Time Frame: Part 2A: 28 days starting from the first 116 or 152 mg dose
Population: All enrolled participants in Part 2A who received the planned 2 doses of 116 mg or 152 mg of study intervention during the DLT observation period or who received at least 1 dose of 116 mg or 152 mg of study intervention and experience DLT(s) during the DLT observation period. Here "Overall Number of Participants Analyzed" signifies the number of participants evaluable for this outcome measure. This outcome measure was not planned to be analyzed in Part 1 and Part 2B of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: Dose Level 1 | Part 2A: Dose Level 2
Number analyzed (Participants) | 7 | 7
Participants | 1 | 1

3. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious AEs (SAEs) [All Causalities and Treatment Related]: Parts 1 and 2
Description: An AE is any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An SAE is defined as any untoward medical occurrence that, at any dose, meets 1 or more of the criteria listed below: Results in death, requires inpatient hospitalization or prolongation of existing hospitalization, life-threatening, congenital anomaly/birth defect etc. A treatment-related AE was any untoward medical occurrence attributed to the study drug in a participant who received study drug. Relatedness to study drug was assessed by the investigator.
Time Frame: Day 1 of dosing up to 90 days post last dose (maximum treatment duration 25 cycles, follow up to 790 days)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 | Part 2A: Dose Level 1 | Part 2A: Dose Level 2 | Part 2B
Number analyzed (Participants) | 33 | 12 | 11 | 29
Participants
  All cause: AE | 33 | 12 | 11 | 29
  All cause: SAE | 23 | 11 | 8 | 21
  Treatment related: AE | 32 | 12 | 11 | 25
  Treatment related: SAE | 17 | 10 | 6 | 5

4. Secondary Outcome: Number of Participants With Maximum Grade 3 or 4 and Grade 5 AEs [All Causalities and Treatment Related] Per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5: Parts 1 and 2
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A treatment-related AE was any untoward medical occurrence attributed to the study drug in a participant who received study drug. Relatedness to study drug was assessed by the investigator. AEs were graded according to NCI CTCAE version 5.0 as Grade 1 indicates Mild AE, Grade 2 indicates Moderate AE, Grade 3 indicates severe AE, and grade 4 indicates life-threatening consequences; urgent intervention indicated. Grade 5 indicates death related to AE.
Time Frame: Day 1 of dosing up to 90 days post last dose (maximum treatment duration 25 cycles, follow up to 790 days)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 | Part 2A: Dose Level 1 | Part 2A: Dose Level 2 | Part 2B
Number analyzed (Participants) | 33 | 12 | 11 | 29
Participants
  All cause: Grades 3/4 | 26 | 9 | 6 | 20
  All cause: Grade 5 | 5 | 2 | 4 | 5
  Treatment related: Grades 3/4 | 23 | 10 | 9 | 16
  Treatment related: Grade 5 | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Adverse Events of Special Interest (AESI)- CRS and Immune Effector Cell-associated Neurotoxicity Syndrome (ICANS) [All Causalities and Treatment Related]: Parts 1 and 2
Description: CRS and ICANS were assessed according to ASTCT criteria. ASTCT for ICANS: Grade 1 [immune effector cell-associated encephalopathy (ICE, overall score range 0-10, higher score = better condition) score 7-9, awakens spontaneously]; Grade 2 [ICE score 3-6, awakens to voice]; Grade 3 [ICE score 0-2, awakens only to tactile stimulus, any clinical seizure that resolves rapidly or non-convulsive seizures on EEG that resolve with intervention, focal/local oedema on neuroimaging]; Grade 4 [ICE 0 (unarousable and unable to perform ICE), Unarousable or requires vigorous or repetitive tactile stimuli to arouse. Stupor or coma, Life-threatening prolonged seizure (>5 min); or repetitive clinical or electrical seizures without return to baseline in between, deep focal motor weakness such as hemiparesis or paraparesis, Diffuse cerebral oedema on neuroimaging; decerebrate or decorticate posturing; or cranial nerve VI (abducens nerve) palsy; or papilledema; or Cushing's triad].
Time Frame: Day 1 of dosing up to 90 days post last dose (maximum treatment duration 25 cycles, follow up to 790 days)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 | Part 2A: Dose Level 1 | Part 2A: Dose Level 2 | Part 2B
Number analyzed (Participants) | 33 | 12 | 11 | 29
Participants
  All cause: CRS | 20 | 10 | 10 | 14
  All cause: ICANS | 1 | 1 | 2 | 0
  Treatment related: CRS | 20 | 10 | 10 | 13
  Treatment related: ICANS | 1 | 1 | 2 | 0

6. Secondary Outcome: Number of Participants With Hematological Measures With Baseline CTCAE Grade >=2 Shifted to a Maximum CTCAE Grade 3-4: Parts 1 and 2
Description: Hematology results were graded according to the NCI CTCAE version 5.0 for relevant parameters, Grade 1 indicates Mild AE, Grade 2 indicates Moderate AE, Grade 3 indicates severe AE, and grade 4 indicates life-threatening consequences; urgent intervention indicated, Grade 5 indicates death related to AE. Hematological measures included Hemoglobin, Platelet count, WBC count, Plasma cell count. Absolute: Neutrophils, Eosinophils, Monocytes, Basophils, Lymphocytes, Plasma cells etc.
Time Frame: Parts 1 and 2: From start of treatment to end of the study (approximately 3 years 7 months)
Reporting Status: Not Posted, anticipated posting 2026-10

7. Secondary Outcome: Number of Participants With Clinical Chemistry Parameters With Baseline CTCAE Grade >=2 Shifted to a Maximum CTCAE Grade 3-4: Parts 1 and 2
Description: Clinical chemistry data included BUN (Blood urea nitrogen), Creatinine, Glucose (non-fasting), Total Calcium, Sodium, Potassium, Chloride, Magnesium, Phosphorus or Phosphates, Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), Total bilirubin, Alkaline phosphatase, Albumin, Chloride, Total CO2 (bicarbonate), Total protein, Lactate dehydrogenase (LDH), Uric acid, Serum beta-2 microglobulin.
Time Frame: Parts 1 and 2: From start of treatment to end of the study (approximately 3 years 7 months)
Reporting Status: Not Posted, anticipated posting 2026-10

8. Secondary Outcome: Number of Participants With Liver Function Tests Abnormalities: Parts 1 and 2
Description: Alanine aminotransferase, aspartate aminotransferase, Alkaline Phosphatase, and total bilirubin (TBILI) were used to assess possible drug induced liver toxicity.
Time Frame: Parts 1 and 2: From start of treatment to end of the study (approximately 3 years 7 months)
Reporting Status: Not Posted, anticipated posting 2026-10

9. Secondary Outcome: Objective Response Rate (ORR) Per International Myeloma Working Group (IMWG) Response Criteria as Determined by Investigator: Parts 1 and 2
Description: ORR: % of participants with objective response. stringent complete response (sCR):CR; ii) normal serum free light chain (FLC) ratio; absence of clonal cells in bone marrow biopsy (BMB)/ bone marrow aspirate (BMA) by immunohistochemistry or immunofluorescence. CR: negative immunofixation on serum and urine, disappearance of any soft tissue plasmacytomas and <5% plasma cells in BMA. If the only measurable disease is by serum FLC levels, CR was normal serum FLC ratio of 0.26-1.65. VGPR:Serum and urine M-protein detectable by immunofixation but not on electrophoresis;>=90% reduction in serum M-protein plus urine M-protein level <100 mg/24 h; if only measurable disease is by serum FLC levels, VGPR:>=90% decrease in difference between involved and uninvolved serum FLC levels; in addition if present at baseline, >90% reduction compared to baseline in size of soft tissue plasmacytomas. PR:≥50% reduction of serum M-protein and reduction in 24 hours urinary M-protein by ≥90% or to <200 mg/24 h.
Time Frame: Parts 1 and 2: From start of treatment to end of the study (approximately 3 years 7 months)
Reporting Status: Not Posted, anticipated posting 2026-10

10. Secondary Outcome: Complete Response Rate (CRR) Per IMWG Response Criteria as Determined by Investigator: Parts 1 and 2
Description: CRR was defined as the percentage of participants with a BOR of confirmed sCR/CR per IMWG response criteria as determined by investigator. sCR: i) CR; ii) normal serum FLC ratio and absence of clonal cells in BMB/BMA by immunohistochemistry or immunofluorescence (κ/λ ratio <=4:1 or >=1:2 for κ and λ participants, respectively, after counting >=100 plasma cells; iii) if the only measurable disease was by serum FLC levels, sCR was defined as normal serum FLC ratio of 0.26 to 1.65 plus absence of clonal cells in BMB/BMA b by immunohistochemistry or immunofluorescence (κ/λ ratio <=4:1 or >=1:2 for κ and λ participants, respectively, after counting >=100 plasma cells). CR: i) negative immunofixation on serum and urine, disappearance of any soft tissue plasmacytomas and <5% plasma cells in BMA; ii) if the only measurable disease was by serum FLC levels, CR was defined as normal serum FLC ratio of 0.26 to 1.65 plus criteria (i).
Time Frame: Parts 1 and 2: From start of treatment to end of the study (approximately 3 years 7 months)
Reporting Status: Not Posted, anticipated posting 2026-10

11. Secondary Outcome: Time to Response (TTR) Per IMWG Response Criteria as Determined by Investigator: Parts 1 and 2
Description: Time to response was defined for participants with an objective response per IMWG criteria, as the time from the date of first dose to the first documentation of objective response that was subsequently confirmed.
Time Frame: Parts 1 and 2: From start of treatment to end of the study (approximately 3 years 7 months)
Reporting Status: Not Posted, anticipated posting 2026-10

12. Secondary Outcome: Duration of Response (DOR) Per IMWG Response Criteria as Determined by Investigator: Parts 1 and 2
Description: DOR: time from the first documentation of objective response, until confirmed PD, or death due to any cause, whichever occurred first. PD: Increase of >=25% from lowest confirmed response value in any 1 or more of following: serum M-component (absolute increase must be >=0.5 g/dL); serum M-protein increase >=1 g/dL, if lowest M component was >=5 g/dL; urine M-protein (absolute increase must be >=200 mg/24 h). In participants without measurable serum and urine M-protein levels, difference between involved and uninvolved serum FLC levels (absolute increase must be >10 mg/dL). In participants without measurable serum, urine M-protein levels and involved serum FLC levels, BM plasma-cell % irrespective of baseline status (must be >=10%). Appearance of a new lesion, >=50% increase from nadir in SPD of >1 lesion, or >=50% increase in longest diameter of a previous lesion >1 cm in short axis. >=50% increase in circulating plasma cells (minimum of 200 cells per mcL) if only measure of disease.
Time Frame: Parts 1 and 2: From start of treatment to end of the study (approximately 3 years 7 months)
Reporting Status: Not Posted, anticipated posting 2026-10

13. Secondary Outcome: Duration of Complete Response Rate (DOCR) Per IMWG Response Criteria as Determined by Investigator: Parts 1 and 2
Description: DOCR was defined as the time from the first documentation of sCR or CR that was subsequently confirmed, until confirmed PD per IMWG criteria, or death due to any cause, whichever occurred first. sCR: i) CR; ii) normal serum FLC ratio and absence of clonal cells in BMB/BMA by immunohistochemistry or immunofluorescence (κ/λ ratio <=4:1 or >=1:2 for κ and λ participants, respectively, after counting >=100 plasma cells; iii) if the only measurable disease was by serum FLC levels, sCR was defined as normal serum FLC ratio of 0.26 to 1.65 plus absence of clonal cells in BMB/BMA b by immunohistochemistry or immunofluorescence (κ/λ ratio <=4:1 or >=1:2 for κ and λ participants, respectively, after counting >=100 plasma cells). CR: i) negative immunofixation on serum and urine, disappearance of any soft tissue plasmacytomas and <5% plasma cells in BMA; ii) if the only measurable disease was by serum FLC levels, CR was defined as normal serum FLC ratio of 0.26 to 1.65 plus criteria (i).
Time Frame: Parts 1 and 2: From start of treatment to end of the study (approximately 3 years 7 months)
Reporting Status: Not Posted, anticipated posting 2026-10

14. Secondary Outcome: Progression Free Survival (PFS) Per IMWG Response Criteria as Determined by Investigator: Parts 1 and 2
Description: PFS was defined as the time from the date of first dose until confirmed PD per IMWG criteria, or death due to any cause, whichever occurred first. Analysis was performed using Kaplan-Meier method. Participants with no PD event or death or who started a new anticancer therapy prior to an event or with an event after a gap of 2 or more missing disease assessments were censored on the date of last adequate disease assessment. Participants who did not have an adequate post-baseline disease assessment were censored on the date of first dose of study intervention unless death occurred on or before the time of the second planned disease assessment (<=8 weeks after the date of first dose) in which case the death was considered an event.
Time Frame: Parts 1 and 2: From start of treatment to end of the study (approximately 3 years 7 months)
Reporting Status: Not Posted, anticipated posting 2026-10

15. Secondary Outcome: Overall Survival (OS): Parts 1 and 2
Description: OS was defined as the time from the date of first dose until death due to any cause. If a participant was not known to have died, survival was censored at the date of last contact. Analysis was performed using Kaplan-Meier method.
Time Frame: Parts 1 and 2: From start of treatment to end of the study (approximately 3 years 7 months)
Reporting Status: Not Posted, anticipated posting 2026-10

16. Secondary Outcome: Minimal Residual Disease (MRD) Negativity Rate Per IMWG Sequencing Criteria: Parts 1 and 2
Description: MRD negativity rate was defined as the percentage of participants with negative MRD (assessed by central laboratory) per IMWG sequencing criteria at any time from the date of first dose until the first documentation of confirmed PD, death or start of new anticancer therapy, whichever occurred first. Sequencing MRD negative included: 1) CR: negative immunofixation on serum and urine, disappearance of any soft tissue plasmacytomas and <5% plasma cells in BMA. If the only measurable disease is by serum FLC levels, CR was defined as normal serum FLC ratio of 0.26 to 1.65; 2) Absence of clonal plasma cells by next generation sequencing (NGS) on BMA in which presence of a clone was defined as <2 identical sequencing reads obtained after DNA sequencing of BMA using the LymphoSIGHT platform (or validated equivalent method) with a minimum sensitivity of 1 in 10^5 nucleated cells.
Time Frame: Parts 1 and 2: From start of treatment to end of the study (approximately 3 years 7 months)
Reporting Status: Not Posted, anticipated posting 2026-10

17. Secondary Outcome: Pre- and Post-dose Concentrations of Elranatamab: Parts 1 and 2
Time Frame: Parts 1 and 2: Till study completion approximately 3 years 7 months
Reporting Status: Not Posted, anticipated posting 2026-10

18. Secondary Outcome: Number of Participants With Anti-Drug Antibody (ADA) and Neutralizing Antibody (Nab) Against Elranatamab: Parts 1 and 2
Time Frame: Parts 1 and 2: From start of treatment to end of the study (approximately 3 years 7 months)
Reporting Status: Not Posted, anticipated posting 2026-10

ADVERSE EVENTS:
Time Frame: Day 1 of dosing up to 90 days post last dose (maximum treatment duration 25 cycles, follow up to 790 days)
Description: Same event may appear as both non-SAE and SAE. What is presented are distinct events. An event may be categorized as serious in 1 participant and non-serious in other participant, or a participant may have experienced both SAE and non-SAE. Safety analysis set evaluated. All-cause mortality: number of deaths are reported from Day 1 of the study up to 90 days post last dose and deaths which occurred after 90 days post last dose of study drug are also included.
Arm/Group | Part 1 | Part 2A: Dose Level 1 | Part 2A: Dose Level 2 | Part 2B
All-Cause Mortality (participants affected / at risk) | 13/33 | 8/12 | 4/11 | 8/29
Serious Adverse Events (participants affected / at risk) | 23/33 | 11/12 | 8/11 | 21/29
Other Adverse Events (participants affected / at risk) | 33/33 | 12/12 | 10/11 | 28/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 (N=33) | Part 2A: Dose Level 1 (N=12) | Part 2A: Dose Level 2 (N=11) | Part 2B (N=29)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Deafness bilateral (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0
Disease progression (General disorders) | 3 | 1 | 2 | 3
Malaise (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 6 | 6 | 3 | 3
Adenovirus infection (Infections and infestations) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 2 | 1 | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 1 | 3 | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 1 | 1
Cytomegalovirus chorioretinitis (Infections and infestations) | 1 | 0 | 0 | 0
Cytomegalovirus infection reactivation (Infections and infestations) | 1 | 0 | 0 | 0
Cytomegalovirus viraemia (Infections and infestations) | 2 | 0 | 0 | 0
Enterovirus infection (Infections and infestations) | 0 | 0 | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0 | 0 | 2
Fungaemia (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 1 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 0 | 3 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia proteus (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia pseudomonal (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia viral (Infections and infestations) | 1 | 0 | 1 | 0
Sepsis (Infections and infestations) | 3 | 1 | 1 | 1
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Soft tissue infection (Infections and infestations) | 1 | 0 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 2 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 0 | 1 | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 (N=33) | Part 2A: Dose Level 1 (N=12) | Part 2A: Dose Level 2 (N=11) | Part 2B (N=29)
Anaemia (Blood and lymphatic system disorders) | 15 | 6 | 5 | 15
Leukopenia (Blood and lymphatic system disorders) | 10 | 4 | 3 | 8
Lymphopenia (Blood and lymphatic system disorders) | 2 | 2 | 3 | 4
Neutropenia (Blood and lymphatic system disorders) | 19 | 7 | 6 | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 6 | 4 | 13
Constipation (Gastrointestinal disorders) | 7 | 1 | 2 | 8
Diarrhoea (Gastrointestinal disorders) | 17 | 6 | 2 | 9
Nausea (Gastrointestinal disorders) | 9 | 4 | 2 | 5
Vomiting (Gastrointestinal disorders) | 6 | 2 | 2 | 4
Fatigue (General disorders) | 13 | 7 | 6 | 13
Influenza like illness (General disorders) | 3 | 2 | 1 | 1
Injection site erythema (General disorders) | 6 | 2 | 3 | 2
Injection site reaction (General disorders) | 10 | 7 | 3 | 8
Malaise (General disorders) | 3 | 1 | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 1 | 1 | 1
Oedema peripheral (General disorders) | 2 | 0 | 3 | 2
Pyrexia (General disorders) | 14 | 4 | 0 | 4
Cytokine release syndrome (Immune system disorders) | 15 | 7 | 8 | 13
Hypogammaglobulinaemia (Immune system disorders) | 12 | 1 | 1 | 3
COVID-19 (Infections and infestations) | 2 | 2 | 0 | 4
Cellulitis (Infections and infestations) | 1 | 1 | 1 | 3
Cytomegalovirus infection reactivation (Infections and infestations) | 4 | 0 | 2 | 3
Cytomegalovirus viraemia (Infections and infestations) | 4 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 4 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 5 | 0 | 0 | 0
Rhinovirus infection (Infections and infestations) | 3 | 1 | 0 | 2
Sinusitis (Infections and infestations) | 4 | 0 | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 6 | 1 | 0 | 2
Viral upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 3
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 2
Alanine aminotransferase increased (Investigations) | 1 | 1 | 1 | 5
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 1 | 2
Blood creatinine increased (Investigations) | 2 | 2 | 3 | 4
Weight decreased (Investigations) | 4 | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 13 | 7 | 3 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 1 | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 5 | 1 | 0 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 2 | 0 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 2 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 5 | 1 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 4 | 1 | 3
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 4
Headache (Nervous system disorders) | 10 | 0 | 2 | 5
Depression (Psychiatric disorders) | 2 | 1 | 1 | 2
Insomnia (Psychiatric disorders) | 3 | 1 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 2 | 1 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 1 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 2 | 4 | 6
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 1 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 3 | 1 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 3
Hypertension (Vascular disorders) | 4 | 0 | 0 | 1
Hypotension (Vascular disorders) | 4 | 1 | 1 | 1

LIMITATIONS AND CAVEATS:
ASTCT: American Society for Transplantation and Cellular Therapy.

CTCAE: Common Terminology Criteria for Adverse Events.

g/dl: Gram/deciliter

mg: Milligram

BM: Bone marrow

Cm: Centimeter

SPD: Sum of the products of diameters

mcl: Microliter

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/12/NCT05014412/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-31): https://cdn.clinicaltrials.gov/large-docs/12/NCT05014412/SAP_001.pdf